CLINICAL TRIAL: NCT00541034
Title: Phase II Study of Pentostatin With Cyclophosphamide and Rituximab for Previously Untreated Patients With Chronic Lymphocytic Leukemia
Brief Title: Pentostatin, Cyclophosphamide, and Rituximab in Treating Patients With Previously Untreated Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-051; P30CA008748 (NIH); MSKCC-05051
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-07

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell chronic lymphocytic leukemia; stage I small lymphocytic lymphoma; stage II small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Cyclophosphamide; Pentostatin

ARMS (1):
- cyclophosphamide, pentostatin & rituximab (Experimental): Patients receive cyclophosphamide IV followed by pentostatin IV on day 1 in course 1. Beginning in course 2 and in all subsequent courses, patients receive cyclophosphamide IV on day 1, pentostatin IV on day 1, and rituximab IV on day 1 or on days 1 and 2. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: pentostatin

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: pentostatin

SUMMARY:
RATIONALE: Pentostatin may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving pentostatin together with cyclophosphamide and rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying the side effects and how well giving pentostatin together with cyclophosphamide and rituximab works in treating patients with previously untreated chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the frequency of response in patients with previously untreated, intermediate- or high-risk B-cell chronic lymphocytic leukemia (CLL) treated with pentostatin, cyclophosphamide, and rituximab.
* To characterize the toxicity of this regimen in these patients.

OUTLINE: Patients receive cyclophosphamide IV followed by pentostatin IV on day 1 in course 1. Beginning in course 2 and in all subsequent courses, patients receive cyclophosphamide IV on day 1, pentostatin IV on day 1, and rituximab IV on day 1 or on days 1 and 2. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at least every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic lymphocytic leukemia (CLL), as evidenced by an absolute lymphocytosis in the blood of at least 5,000 lymphocytes per microliter OR bone marrow lymphocytosis ≥ 30% of all nucleated cells

  * Previously untreated disease
* Meets 1 of the following risk criteria as defined by the three-stage Rai system

  * Intermediate-risk disease

    * Must meet the criteria for active disease as defined by the NCI Working Group guidelines including the following:

      * Weight loss
      * Fatigue
      * Fevers
      * Evidence of progressive marrow failure
      * Splenomegaly
      * Progressive lymphadenopathy
      * Progressive lymphocytosis with a rapid doubling time
  * High-risk disease
* Malignant lymphocytes must demonstrate B-cells via immunophenotypic or immunohistochemical analysis
* Patients with small lymphocytic lymphoma (CLL type) are eligible

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status 60-100%
* Total bilirubin ≤ 2.0 mg/dL (patients with Gilbert disease or autoimmune hemolytic anemia should have an evaluation for other causes of hyperbilirubinemia, but if none are found they may be enrolled regardless of serum bilirubin)
* Total creatinine ≤ 2.0 mg/dL OR creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Patients with autoimmune hemolytic anemia or autoimmune thrombocytopenia are eligible for treatment on this protocol regardless of disease stage

Exclusion criteria:

* Significant active infections
* Ongoing hepatitis B infection, specifically hepatitis B antigen or surface antigen positivity

  * Patients who are hepatitis B antibody positive are eligible for this protocol

PRIOR CONCURRENT THERAPY:

* Concurrent prednisone allowed provided it is used as brief courses (≤ 7 days) for inflammatory conditions unrelated to CLL
* No prior cytotoxic therapy or rituximab for this cancer
* No concurrent radiotherapy or other chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Lamanna, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Renier Brentjens, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients who received cyclophosphamide, pentostatin and rituximab
Period: Overall Study
Arm/Group | All Patients
Started | 49
Completed | 46
Not Completed | 3
Not completed — Non-Compliance | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: The major criteria for determination of response to therapy in patients with CLL include physical examination and examination of the peripheral blood and bone marrow. Radiographic studies are not required but those that were abnormal pre-treatment, will be repeated to document the degree of maximal response.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 46
Participants
  Complete Response (CR) | 10
  Nodular Response | 5
  Partial Response (PR) | 26
  Stable Disease (SD) | 4
  Progression of Disease (POD) | 1

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 18/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=49)
Dizziness (General disorders) | 1
Dyspnea (General disorders) | 3
Facial pain (General disorders) | 1
Febrile neutropenia (General disorders) | 5
Hypertension (Cardiac disorders) | 2
Immune system disorder (Immune system disorders) | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1
Localized edema (General disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Pharyngeal mucositis (General disorders) | 1
Pneumonia (General disorders) | 9
Rash desquamating (Skin and subcutaneous tissue disorders) | 1
Tooth infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=49)
ALT, SGPT (Blood and lymphatic system disorders) | 9
AST, SGOT (Blood and lymphatic system disorders) | 4
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 9
Creatinine (Metabolism and nutrition disorders) | 3
Distension/bloating, abdominal (Gastrointestinal disorders) | 3
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 32
Hemoglobin (Blood and lymphatic system disorders) | 42
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 39
Lymphopenia (Blood and lymphatic system disorders) | 31
Nausea (Gastrointestinal disorders) | 4
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 46
Pain (General disorders) | 3
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 13
Platelets (Blood and lymphatic system disorders) | 21
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 7
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 3
Tumor lysis syndrome (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes